CLINICAL TRIAL: NCT03338595
Title: Longitudinal Assessment of Exercise Capacity and Vascular Function in Patients With CF
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Principal Investigator, Ryan Harris, Principal Investigator, Augusta University
Other Study IDs: CF-Long
Record Dates: First submitted 2017-03-31; First posted 2017-11-09 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Cystic Fibrosis
Keywords: arterial stiffness; flow-mediated dilation; endothelial function; Orkambi; exercise capacity
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project is an attempt to understand how Orkambi treatment affects exercise capacity and the function of the arteries in CF patients who are homozygous F508del. Our goal is to perform the exercise and vascular measurements every 3 months after a patient starts taking Orkambi.

DETAILED DESCRIPTION:
Cystic Fibrosis (CF) is the most common fatal genetic disease in North America. The most disturbing aspect of CF is the associated premature death, most often due to respiratory complications. Clinical manifestations of CF include not only lung dysfunction, but many other systemic consequences as well. Systemic oxidative stress and exercise intolerance are established phenotypes in patients with CF. Additionally, for the first time the investigators have recently published the presence of systemic endothelial dysfunction in a cohort of young patients with CF who exhibited normal oxygen saturation and spirometric function.

Exercise intolerance, the limitation of the ability to perform exercise at the expected level, has been shown to predict mortality in patients with CF independent of lung function. Exercise capacity (VO2 peak), an objective measurement of exercise tolerance, drops approximately 5-8% per year in patients with CF. This excessive decay in exercise capacity not only leads to more pulmonary infections and deterioration of lung function, it represents a 5-8 fold decline compared to healthy sedentary adults. Preventing the excessive annual reduction in exercise capacity is essential to increasing the quality of life and longevity of patients with CF. However, a critical barrier to improving exercise capacity in CF is the investigators lack of knowledge regarding the different physiological mechanisms that contribute to exercise intolerance. It is important to emphasize that decreases in lung function (FEV1) do not always contribute to reductions in VO2 peak. Furthermore, less than 2% of patients who have an FEV1 greater than 50% predicted will have a significant drop in hemoglobin oxygen saturation (SpO2) during maximal exercise. These data suggest that mechanisms other than lung function induced hypoxemia may be contributing to exercise intolerance in patients with CF.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Cystic Fibrosis (homozygous deltaF508del)
* Prescribed Orkambi
* Men and women (> 18 yrs. old)
* Boys and girls (7 -17 yrs. old)
* FEV1 percent predicted > 40%
* Resting oxygen saturation (room air) >85%
* Patients with or without CFRD
* Traditional CF-treatment medications
* Clinically stable for past 28 days (no exacerbations or change in medical status)
* Healthy Controls

Exclusion Criteria:

* Children 6 yrs. old and younger
* FEV1 percent predicted < 40%
* Resting oxygen saturation (room air) < 85%
* Clinical diagnosis of heart disease
* Pulmonary artery hypertension
* Febrile illness within two weeks of visit
* Current smokers
* Currently pregnant or nursing
* Individuals on vaso-active medications (i.e. nitrates, beta blockers, ACE inhibitors, etc.)
* Use of VX-770 within 6 months prior to Visit 1
* History of solid organ transplantation
* Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or the quality of the data.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: CF patients who are homozygous F508del and have been prescribed Orkambi.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Maximal exercise capacity | 1 year
  Subjects will perform the maximal exercise tests on an electronically braked cycle ergometer using the Godfrey protocol. Expired gases will be collected using a Parvo Medics True One metabolic cart for determination of exercise capacity (VO2 peak).

SECONDARY OUTCOMES:
Flow mediated dilation | 1 year
  The brachial artery FMD test will be performed according to the recent tutorial on the ultrasonic assessment of FMD and shear rate will be calculated as the stimulus of the vasodilatory response. Briefly, subjects will lie in the supine position for 20 minutes to obtain hemodynamic steady state. A blood pressure cuff (Hokanson) will be placed around the forearm (distal to the Doppler transducer) and rapidly inflated to 250 mmHg for 5 minutes (circulatory arrest). Simultaneous ultrasound images of the vessel (B-mode) and Doppler waveforms will be collected 10 seconds prior to and for 2 minutes following deflation of the cuff.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Harris, PhD, Principal Investigator — Augusta University
Locations (1):
- Georgia Prevention Institute, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes